CLINICAL TRIAL: NCT01591616
Title: A Phase 4 Pediatric Study to Assess the Pharmacokinetics and Safety of Oraqix Gel in Healthy Children and Adolescent Volunteers Following Tooth Extraction
Brief Title: Pediatric Study to Access Pharmacokinetics and Safety of Oraqix Gel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Dentsply International (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TP73
Record Dates: First submitted 2011-06-24; First posted 2012-05-04 (Estimated); Results first posted 2014-04-03 (Estimated); Last update posted 2020-08-07 (Actual); Status verified 2020-07

CONDITIONS: Periodontal Disease
MeSH Terms: conditions — Periodontal Diseases | interventions — Lidocaine, Prilocaine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oraqix for tooth extraction (Other)
  Interventions: Drug: lidocaine and prilocaine

INTERVENTIONS:
Drug: lidocaine and prilocaine — Appropriate dose of Oraqix based on weight will be given before tooth extraction
  Other Names: Oraqix periodontal gel

SUMMARY:
To establish Oraqix is safe when used on adolescent volunteers.

DETAILED DESCRIPTION:
This is a single-center, uncontrolled, open-label, single administration patient study. Male and female subjects aged 6 through 17 years of age in need of primary tooth extraction will be recruited from the Principal Investigator's database and may be supplemented by advertising. Subjects who withdraw from the study prematurely will be replaced.

Subjects will undergo an initial screening visit at which eligibility will be determined. After completion of informed consent/assent a physical examination, vitals, 12-lead ECG, and dental examination will be conducted. A medical history will be documented and a blood sample will be collected for analysis of biochemistry, hematology and as appropriate, serum pregnancy assessment for females.

Subjects will return to the office approximately 1 to 10 days after Visit 1 for Visit 2. At Visit 2, study treatment will be administered and PK blood samples will be collected for analysis, and monitored for safety parameters. Up to a total of five cartridges of Oraqix® will be administered to the oral cavity in the area of the tooth extraction, based on the body weight of the subject. No more than five cartridges will be dispensed, since this is the maximum dose for this agent. The final sample will be collected 4 hours after administration of study material. An abbreviated dental examination will be conducted, any adverse events (AEs) will be documented and the subject will be discharged from the clinic.

All subjects will be contacted by telephone approximately 24 hours after administration of study treatment. Study personnel will enquire about the occurrence of any AEs that have occurred since leaving the office. If appropriate, further follow-up of AEs will be arranged. In the absence of any ongoing AEs requiring follow up the subject will be considered to have completed the study at the completion of the telephone call.

ELIGIBILITY:
Inclusion Criteria:

* 6 and 17 and eleven twelfths
* requires tooth extraction
* healthy having not taken any prescription or over the counter medications within 60 days of first visit
* must be a minimum of 15 kg

Exclusion Criteria:

* anesthesia required for treatment other than study material
* given blood within 90 days of first visit
* pregnant
* allergic to local anesthetic
* documented history of glucose-6-phosphate dehydrogenase deficiency
* history of congenital idiopathic methemoglobinemia
* does not have a loose tooth easily extracted or who, in the opinion of the Investigator, is not suitable for tooth extraction using only topical anesthetic

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 16 (Actual)
Dates: Start 2010-04; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tegwyn Brickhouse, D.D.S PhD, Principal Investigator — Virginia Commonweath School of Dentistry
Locations (1):
- Virginia Commonweath School of Dentistry, Richmond, Virginia, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Oraqix for Tooth Extraction
Started | 16
Completed | 15
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Oraqix for Tooth Extraction
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 16
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 7
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Pharmacokinetics
Description: The study focused on the pharmacokinetics of prilocaine and lidocaine, o-toluidine (metabolite of prilocaine) and 2, 6-xylidine (metabolite of lidocaine). We evaluated blood samples of15 subjects at the following time points: pre-dose, at 5,10,15,30, 60, 90, 120 and 240 min post dose. We calculated Cmax (maximum observed plasma concentration) and Tmax (time to maximum plasma concentration).
Time Frame: 5, 10, 15, 30, 60, 90, 120, and 240 minutes
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Lidocaine Cmax | Prilocaine Cmax | 2,6-xylidine Cmax | O-toluidine Cmax
Number analyzed (Participants) | 15 | 15 | 11 | 15
ng/mL | 89.9 (66) | 41.8 (60.6) | 3.72 (48.5) | 5.13 (51.2)

2. Secondary Outcome: Safety
Description: The % MetHb levels and vital signs (pulse, systolic and diastolic pressure) were measured at pre-dose (-20, -10 and 0 min prior to Oraqix administration) and every 10 minutes up to 240 minutes post dose.
  ECG taken at pre-dose and 1, 2 and 4h post dose, measurement of heart rate and PR, QRS, QT and QTcB intervals.
  Visual analogue scale conducted at pre-dose (immediately before Oraqix administration), immed. post extraction, at 0.25, 0.5, 1 and 2h post dose and prior to discharge just after 4h post dose.
  For each subject, phone call was made at +24h as follow up pursuant to the protocol.
Time Frame: blood draws pre-dose, 2 and 4 hours postdose
Measure: Mean (Standard Deviation); unit: Percentage MetHb
Groups:
- % MetHemoglobin (MetHb) Time Point -20 Minutes; % MetHemoglobin (MetHb) Time Point -10 Minutes; % MetHemoglobin (MetHb) Time Point 0 Minutes; % MetHemoglobin (MetHb) Time Point 10 Minutes; % MetHemoglobin (MetHb) Time Point 20 Minutes; % MetHemoglobin (MetHb) Time Point 30 Minutes; % MetHemoglobin (MetHb) Time Point 40 Minutes; % MetHemoglobin (MetHb) Time Point 50 Minutes; % MetHemoglobin (MetHb) Time Point 60 Minutes; % MetHemoglobin (MetHb) Time Point 70 Minutes; % MetHemoglobin (MetHb) Time Point 80 Minutes; % MetHemoglobin (MetHb) Time Point 90 Minutes; % MetHemoglobin (MetHb) Time Point 100 Minutes; % MetHemoglobin (MetHb) Time Point 110 Minutes; % MetHemoglobin (MetHb) Time Point 120 Minutes; % MetHemoglobin (MetHb) Time Point 130 Minutes; % MetHemoglobin (MetHb) Time Point 140 Minutes; % MetHemoglobin (MetHb) Time Point 150 Minutes; % MetHemoglobin (MetHb) Time Point 160 Minutes; % MetHemoglobin (MetHb) Time Point 170 Minutes; % MetHemoglobin (MetHb) Time Point 180 Minutes; % MetHemoglobin (MetHb) Time Point 190 Minutes; % MetHemoglobin (MetHb) Time Point 200 Minutes; % MetHemoglobin (MetHb) Time Point 210 Minutes; % MetHemoglobin (MetHb) Time Point 220 Minutes; % MetHemoglobin (MetHb) Time Point 230 Minutes; % MetHemoglobin (MetHb) Time Point 240 Minutes: The % MetHb levels were measured at pre-dose (-20, -10 and 0 min prior to Oraqix administration) and every 10 minutes up to 240 minutes post dose.
Arm/Group | % MetHemoglobin (MetHb) Time Point -20 Minutes | % MetHemoglobin (MetHb) Time Point -10 Minutes | % MetHemoglobin (MetHb) Time Point 0 Minutes | % MetHemoglobin (MetHb) Time Point 10 Minutes | % MetHemoglobin (MetHb) Time Point 20 Minutes | % MetHemoglobin (MetHb) Time Point 30 Minutes | % MetHemoglobin (MetHb) Time Point 40 Minutes | % MetHemoglobin (MetHb) Time Point 50 Minutes | % MetHemoglobin (MetHb) Time Point 60 Minutes | % MetHemoglobin (MetHb) Time Point 70 Minutes | % MetHemoglobin (MetHb) Time Point 80 Minutes | % MetHemoglobin (MetHb) Time Point 90 Minutes | % MetHemoglobin (MetHb) Time Point 100 Minutes | % MetHemoglobin (MetHb) Time Point 110 Minutes | % MetHemoglobin (MetHb) Time Point 120 Minutes | % MetHemoglobin (MetHb) Time Point 130 Minutes | % MetHemoglobin (MetHb) Time Point 140 Minutes | % MetHemoglobin (MetHb) Time Point 150 Minutes | % MetHemoglobin (MetHb) Time Point 160 Minutes | % MetHemoglobin (MetHb) Time Point 170 Minutes | % MetHemoglobin (MetHb) Time Point 180 Minutes | % MetHemoglobin (MetHb) Time Point 190 Minutes | % MetHemoglobin (MetHb) Time Point 200 Minutes | % MetHemoglobin (MetHb) Time Point 210 Minutes | % MetHemoglobin (MetHb) Time Point 220 Minutes | % MetHemoglobin (MetHb) Time Point 230 Minutes | % MetHemoglobin (MetHb) Time Point 240 Minutes
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 15 | 15 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
Percentage MetHb | 1.3 (0.24) | 1.3 (0.26) | 1.2 (0.20) | 1.2 (0.20) | 1.3 (0.18) | 1.5 (0.43) | 1.5 (0.20) | 1.6 (0.19) | 1.7 (0.28) | 1.7 (0.30) | 1.5 (0.35) | 1.5 (0.40) | 1.5 (0.39) | 1.6 (0.19) | 1.5 (0.32) | 1.5 (0.29) | 1.4 (0.28) | 1.4 (0.26) | 1.3 (0.34) | 1.2 (0.47) | 1.4 (0.15) | 1.4 (0.17) | 1.5 (0.20) | 1.4 (0.18) | 1.4 (0.13) | 1.5 (0.14) | 1.4 (0.15)

3. Primary Outcome: Pharmacokinetics
Description: as for outcome 1
Time Frame: 5, 10, 15, 30, 60, 90, 120, and 240 minutes
Measure: Geometric Mean (Full Range); unit: hours
Arm/Group | Lidocaine Tmax | Prilocaine Tmax | 2,6-xylidine Tmax | O-toluidine Tmax
Number analyzed (Participants) | 15 | 15 | 11 | 15
hours | 0.500 [0.0833 to 0.650] | 0.500 [0.0833 to 0.650] | 1.50 [0.650 to 4.00] | 1.50 [1.00 to 1.50]

4. Secondary Outcome: Vital Signs (Pulse)
Description: Vital signs (pulse, systolic and diastolic pressure) were measured at pre-dose (-20, -10 and 0 min prior to Oraqix administration) and every 10 minutes up to 240 minutes post dose.
Time Frame: Pre-dose and every 10 minute to 240 minutes post-dose.
Measure: Mean (Full Range); unit: Beats per minute
Arm/Group | Vital Signs (Pulse Rate), - 20 Minutes Pre-dose | Vital Signs (Pulse Rate), - 10 Minutes Pre-dose | Vital Signs (Pulse Rate), 0 Minutes Pre-dose | Vital Signs (Pulse Rate), 10 Minutes Post-dose | Vital Signs (Pulse Rate), 20 Minutes Post-dose | Vital Signs (Pulse Rate), 30 Minutes Post-dose | Vital Signs (Pulse Rate), 40 Minutes Post-dose | Vital Signs (Pulse Rate), 50 Minutes Post-dose | Vital Signs (Pulse Rate), 60 Minutes Post-dose | Vital Signs (Pulse Rate), 70 Minutes Post-dose | Vital Signs (Pulse Rate), 80 Minutes Post-dose | Vital Signs (Pulse Rate), 90 Minutes Post-dose | Vital Signs (Pulse Rate), 100 Minutes Post-dose | Vital Signs (Pulse Rate), 110 Minutes Post-dose | Vital Signs (Pulse Rate), 120 Minutes Post-dose | Vital Signs (Pulse Rate), 130 Minutes Post-dose | Vital Signs (Pulse Rate), 140 Minutes Post-dose | Vital Signs (Pulse Rate), 150 Minutes Post-dose | Vital Signs (Pulse Rate), 160 Minutes Post-dose | Vital Signs (Pulse Rate), 170 Minutes Post-dose | Vital Signs (Pulse Rate), 180 Minutes Post-dose | Vital Signs (Pulse Rate), 190 Minutes Post-dose | Vital Signs (Pulse Rate), 200 Minutes Post-dose | Vital Signs (Pulse Rate), 210 Minutes Post-dose | Vital Signs (Pulse Rate), 220 Minutes Post-dose | Vital Signs (Pulse Rate), 230 Minutes Post-dose | Vital Signs (Pulse Rate), 240 Minutes Post-dose
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 14 | 14 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
Beats per minute | 74 [58 to 98] | 72 [54 to 90] | 72 [60 to 95] | 79 [59 to 101] | 71 [58 to 89] | 72 [56 to 94] | 71 [55 to 86] | 70 [54 to 86] | 71 [55 to 86] | 74 [61 to 89] | 72 [57 to 86] | 71 [53 to 90] | 70 [54 to 91] | 72 [57 to 88] | 70 [52 to 86] | 71 [58 to 91] | 72 [53 to 97] | 72 [55 to 98] | 74 [58 to 93] | 74 [57 to 100] | 73 [53 to 91] | 72 [50 to 90] | 75 [62 to 90] | 72 [54 to 97] | 70 [53 to 96] | 72 [57 to 96] | 77 [62 to 101]

5. Secondary Outcome: Vital Signs (Systolic Pressure)
Time Frame: Pre-dose (-20, -10 and 0 min prior to Oraqix administration) and every 10 minutes up to 240 minutes post dose.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vital Signs (Systolic), - 20 Minutes Pre-dose | Vital Signs (Systolic), - 10 Minutes Pre-dose | Vital Signs (Systolic), 0 Minutes Pre-dose | Vital Signs (Systolic), 10 Minutes Post-dose | Vital Signs (Systolic), 20 Minutes Post-dose | Vital Signs (Systolic), 30 Minutes Post-dose | Vital Signs (Systolic), 40 Minutes Post-dose | Vital Signs (Systolic), 50 Minutes Post-dose | Vital Signs (Systolic), 60 Minutes Post-dose | Vital Signs (Systolic), 70 Minutes Post-dose | Vital Signs (Systolic) 80 Minutes Post-dose | Vital Signs (Systolic), 90 Minutes Post-dose | Vital Signs (Systolic), 100 Minutes Post-dose | Vital Signs (Systolic), 110 Minutes Post-dose | Vital Signs (Systolic), 120 Minutes Post-dose | Vital Signs (Systolic), 130 Minutes Post-dose | Vital Signs (Systolic), 140 Minutes Post-dose | Vital Signs (Systolic), 150 Minutes Post-dose | Vital Signs (Systolic), 160 Minutes Post-dose | Vital Signs (Systolic), 170 Minutes Post-dose | Vital Signs (Systolic), 180 Minutes Post-dose | Vital Signs (Systolic), 190 Minutes Post-dose | Vital Signs (Systolic), 200 Minutes Post-dose | Vital Signs (Systolic), 210 Minutes Post-dose | Vital Signs (Systolic), 220 Minutes Post-dose | Vital Signs (Systolic), 230 Minutes Post-dose | Vital Signs (Systolic), 240 Minutes Post-dose
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 14 | 14 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
mmHg | 110 (11.5) | 104 (9.4) | 106 (9.1) | 115 (9.7) | 109 (7.9) | 108 (9.4) | 106 (9.8) | 106 (9.6) | 105 (12.1) | 106 (7.9) | 104 (11.0) | 106 (9.7) | 106 (9.9) | 106 (10.7) | 106 (11.4) | 105 (8.9) | 108 (8.0) | 107 (8.4) | 105 (10.7) | 106 (9.6) | 104 (10.2) | 103 (10.7) | 103 (10.9) | 102 (9.2) | 104 (10.8) | 102 (10.6) | 102 (11.7)

6. Secondary Outcome: Vital Signs (Diastolic Pressure)
Time Frame: Pre-dose (-20, -10 and 0 min prior to Oraqix administration) and every 10 minutes up to 240 minutes post dose
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Vital Signs (Diastolic), - 20 Minutes Pre-dose | Vital Signs (Diastolic), - 10 Minutes Pre-dose | Vital Signs (Diastolic), 0 Minutes Pre-dose | Vital Signs (Diastolic), 10 Minutes Post-dose | Vital Signs (Diastolic), 20 Minutes Post-dose | Vital Signs (Diastolic), 30 Minutes Post-dose | Vital Signs (Diastolic), 40 Minutes Post-dose | Vital Signs (Diastolic), 50 Minutes Post-dose | Vital Signs Diastolic(), 60 Minutes Post-dose | Vital Signs (Diastolic), 70 Minutes Post-dose | Vital Signs (Diastolic) 80 Minutes Post-dose | Vital Signs (Diastolic), 90 Minutes Post-dose | Vital Signs (Diastolic), 100 Minutes Post-dose | Vital Signs (Diastolic), 110 Minutes Post-dose | Vital Signs (Diastolic), 120 Minutes Post-dose | Vital Signs Diastolic(), 130 Minutes Post-dose | Vital Signs (Diastolic), 140 Minutes Post-dose | Vital Signs (Diastolic), 150 Minutes Post-dose | Vital Signs (Diastolic), 160 Minutes Post-dose | Vital Signs (Diastolic), 170 Minutes Post-dose | Vital Signs (Diastolic), 180 Minutes Post-dose | Vital Signs (Diastolic), 190 Minutes Post-dose | Vital Signs (Diastolic), 200 Minutes Post-dose | Vital Signs (Diastolic), 210 Minutes Post-dose | Vital Signs (Diastolic), 220 Minutes Post-dose | Vital Signs (Diastolic), 230 Minutes Post-dose | Vital Signs (Diastolic), 240 Minutes Post-dose
Number analyzed (Participants) | 16 | 16 | 16 | 15 | 14 | 14 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 16 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15 | 15
mmHg | 63 (6.8) | 60 (7.2) | 63 (7.2) | 69 (7.9) | 63 (6.2) | 64 (5.6) | 62 (8.7) | 62 (11.2) | 62 (7.7) | 62 (10.8) | 62 (9.3) | 64 (7.6) | 63 (7.6) | 63 (11.4) | 60 (7.6) | 62 (7.9) | 62 (7.2) | 63 (9.1) | 63 (6.6) | 60 (6.8) | 60 (8.8) | 61 (7.1) | 60 (7.6) | 59 (7.5) | 57 (6.9) | 57 (6.9) | 60 (8.4)

7. Secondary Outcome: ECGs (Ventricular Heart Rate)
Description: Ventricular heart rate, PR interval, QRS duration, QT interval, and QTcB intervals were calculated.
Time Frame: Pre-dose, 1 hour, 2 hour, 4 hour post-dose.
Measure: Mean (Standard Deviation); unit: Beats per minute
Arm/Group | Ventricular Heart Rate, Pre-dose | Ventricular Heart Rate, 1 Hour Post-dose | Ventricular Heart Rate, 2 Hour Post-dose | Ventricular Heart Rate, 4 Hour Post-dose
Number analyzed (Participants) | 15 | 15 | 15 | 16
Beats per minute | 73 (9.9) | 70 (8.3) | 71 (6.5) | 74 (10.1)

8. Secondary Outcome: ECGs (PR Interval)
Description: Ventricular heart rate, PR interval, QRS duration, QT interval, and QTcB intervals were calculated.
Time Frame: Pre-dose, 1 hour, 2 hour, 4 hour post-dose.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | PR Interval, Pre-dose | PR Interval, 1 Hour Post-dose | PR Interval, 2 Hour Post-dose | PR Interval, 4 Hour Post-dose
Number analyzed (Participants) | 15 | 15 | 15 | 16
milliseconds | 148 (21.1) | 147 (23.7) | 147 (22.4) | 139 (18.9)

9. Secondary Outcome: ECGs (QRS Duration)
Description: Ventricular heart rate, PR interval, QRS duration, QT interval, and QTcB intervals were calculated.
Time Frame: Pre-dose, 1 hour, 2 hour, 4 hour post-dose.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | QRS Duration, Pre-dose | QRS Duration, 1 Hour Post-dose | QRS Duration, 2 Hour Post-dose | QRS Duration, 4 Hour Post-dose
Number analyzed (Participants) | 15 | 15 | 15 | 16
milliseconds | 77 (5.7) | 76 (4.5) | 75 (7.5) | 74 (5.3)

10. Secondary Outcome: ECGs (QT Interval)
Description: Ventricular heart rate, PR interval, QRS duration, QT interval, and QTcB intervals were calculated.
Time Frame: Pre-dose, 1 hour, 2 hour, 4 hour post-dose.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | QT Interval, Pre-dose | QT Interval, 1 Hour Post-dose | QT Interval, 2 Hour Post-dose | QT Interval, 4 Hour Post-dose
Number analyzed (Participants) | 15 | 15 | 15 | 16
milliseconds | 376 (22.5) | 384 (19.3) | 383 (19.0) | 379 (25.8)

11. Secondary Outcome: ECGs (QTcB Interval)
Description: Ventricular heart rate, PR interval, QRS duration, QT interval, and QTcB intervals were calculated.
Time Frame: Pre-dose, 1 hour, 2 hour, 4 hour post-dose.
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | QTcB Interval, Pre-dose | QTcB Interval, 1 Hour Post-dose | QTcB Interval, 2 Hour Post-dose | QTcB Interval, 4 Hour Post-dose
Number analyzed (Participants) | 15 | 15 | 15 | 16
milliseconds | 412 (19.0) | 413 (21.9) | 415 (18.6) | 419 (21.1)

ADVERSE EVENTS:
Arm/Group | Adverse Events
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 2/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adverse Events (N=16)
Nausea (Gastrointestinal disorders) | 2
Gagging (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Tooth pain (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The subject study was a post-approval requirement related to the approval of NDA 21-451 to evaluate the pharmacokinetics and safety of the Oraqix gel in pediatric patients. As the purpose of the study was solely to fulfill a post approval regulatory requirement, the information is considered proprietary to the sponsor (Dentsply International, Inc.) and disclosure by the Investigators to any third party (unless such disclosure was required by government regulations or laws) was prohibited.